CLINICAL TRIAL: NCT05824494
Title: A Single-arm, Open-label, Multicenter Phase II Study of Cadonilimab Combined With Nab -Paclitaxel in Patients With Persistent, Recurrent, or Metastatic Cervical Cancer Previously Treated With Immune Checkpoint Inhibitors
Brief Title: Cadonilimab Plus Nab -Paclitaxel for Patients With Recurrent, or Metastatic Cervical Cancer Resistant to Immune Checkpoint Inhibitors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-024
Record Dates: First submitted 2023-04-09; First posted 2023-04-21 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Uterine Cervical Neoplasms; Cancer of Cervix; Cervical Cancer; Cervical Neoplasms; Uterine Cervical Cancer; Cancer of the Uterine Cervix
Keywords: PD-1; immune checkpoint inhibitor
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Taxes

STUDY DESIGN:
Intervention Model Description: cadonilimab 10mg/kg Q3W and nab-paclitaxel ≤260mg/m2 Q3W
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab plus nab-paclitaxel (Experimental): Drug: Cadonilimab 10mg/kg,every 3 weeks,IV infusion
  Drug: Nab paclitaxel
  ≤260mg/m2,every 3 weeks,IV infusion
  Interventions: Drug: Cadonilimab; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Cadonilimab — Cadonilimab 10mg/kg,every 3 weeks,IV infusion
Drug: Nab paclitaxel — Nab paclitaxel ≤260mg/m2,every 3 weeks,IV infusion

SUMMARY:
This is a phase II trial of combination therapy of cadonilimab(Bispecific Anti-PD-1/CTLA-4 Antibody) plus nab-Paclitaxel in patients with recurrent or metastatic cervical cancer that had failed PD-1/PD-L1 blockade therapy. As a bispecific antibody against PD-1 and CTLA-4, cardonirimab can not only induce the production of a large number of T cells in the early stage of immune response by antagonizing CTLA-4, but also block PD-1 and PD-L1/L2 combination. Thereby restoring the killing function of T cells to tumor cells and reducing the exhaustion of T cells.The hypothesis is the combination of cadonilimab and nab-Paclitaxel will overcome PD-1/PD-L1 blockade-resistance to enhance the response of patients with persistant, recurrent or metastatic cervical cancer.

DETAILED DESCRIPTION:
Primary objective:

Objective response rate for cadonilimab in combination with nab-paclitaxel in the treatment of persistent, recurrent, or metastatic cervical cancer previously treated with immune checkpoint inhibitors.

Secondary objective:

To evaluate duration of response (DoR) and disease control rate (DCR) of cardinirimab combined with nab-paclitaxel in the treatment of persistent, recurrent or metastatic cervical cancer who have previously received immune checkpoint inhibitor therapy based on RECIST v1.1 and time to response (TTR).

To evaluate the progression-free survival (PFS) and overall survival (OS) of patients with persistent, recurrent or metastatic cervical cancer who had previously received immune checkpoint inhibitor therapy with cardonilimab combined with nab-paclitaxel.

To evaluate the safety and tolerability of this combination therapy.

Exploratory objective:

To search for potential indicators in tumor tissue or peripheral blood of subjects that can predict the efficacy of cardonirimab combined with nab-paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are autonomous and fully autonomous, understand and voluntarily sign a written informed consent within 30 days before enrollment.
2. Age ≥ 18 and ≤ 75 years old on the date of signing the informed consent form, female.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
4. Expected survival period ≥ 3 months.
5. Persistent, recurrent or metastatic cervical cancer confirmed by histology or cytology.
6. Subjects who have previously failed treatment with PD-1, PD-L1 or CTLA4 inhibitors.
7. There is at least one measurable tumor lesion according to the RECIST v1.1 standard; tumor lesions in the previous radiotherapy area or other locoregional treatment sites are generally not regarded as measurable lesions, unless the lesion has definite progression and persists after 3 months of radiotherapy, Or the tumor nature of the lesion is confirmed by biopsy.
8. All subjects need to provide informed consent to provide freshly obtained tumor tissue samples or tumor tissue samples archived within 5 years (formalin-fixed paraffin-embedded [FFPE] tissue wax blocks or at least 5 unstained tumor tissue Biopsy samples, preferably freshly obtained tumor tissue samples). If the subject cannot provide the tumor tissue sample archived within 5 years before randomization or the tumor tissue sample is not suitable for use, a biopsy must be performed to collect fresh tumor tissue; if the investigator judges that there is a safety risk in the subject's tumor tissue biopsy, the Discuss with medical monitor.
9. The subject agrees to collect tumor tissue and peripheral blood samples required during the screening period and the research process and apply them to relevant research.
10. The results of laboratory tests after the screening period suggest that the subject has good organ function:

    1. Hematology (no blood components and cell growth factor supportive treatment are allowed within 2 weeks before randomization): i. The absolute value of neutrophils ANC ≥ 1.5 × 109/L (1,500/mm3); ii. Platelet count ≥ 100 × 109/L (100,000/mm3); iii. Hemoglobin ≥ 90 g/L.
    2. Kidneys: i. Calculated creatinine clearance* (CrCl) ≥ 50 mL/min

       * CrCl will be calculated using the Cockcroft-Gault formula (Cockcroft-Gault formula) CrCl (mL/min) = {(140 - age) × body weight (kg) × 0.85}/ (serum creatinine. (mg/dL) × 72) ii. Urinary protein < 2+ or 24-hour (h) urine protein quantitative < 1.0 g.
    3. Liver: i. Serum total bilirubin (TBil) ≤ 1.5 × ULN ii. AST and ALT ≤ 2.5× ULN iii. Serum albumin (ALB) ≥ 28 g/L
    4. coagulation function: i. International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (if the subject is receiving anticoagulant therapy, the subject must receive a stable dose of anticoagulant and coagulation parameters at the time of screening (PT/INR and APTT) were within expected ranges with anticoagulant therapy).
    5. Cardiac function: i. Left ventricular ejection fraction (LVEF) ≥ 50%.
11. Female subjects of childbearing potential must have a serum pregnancy test within 3 days before the first dose and the result is negative. If a female subject of childbearing potential has sex with an unsterilized male partner, the subject must use an acceptable and effective method of contraception since screening and must agree to continue using these precautions until after the last dose of the study drug 6 months; Periodic abstinence and rhythm contraception are unacceptable contraceptive methods.

    1. Females of childbearing potential are defined as females who have not been surgically sterilized (i.e. bilateral tubal ligation, bilateral oophorectomy, or total hysterectomy) or who have not undergone menopause (menopause is defined as at least Menopause for 12 consecutive months, serum follicle-stimulating hormone level is within the laboratory reference range for postmenopausal women);
    2. A highly effective contraceptive method is one that has a low rate of contraceptive failure (eg, less than 1% per year) when used correctly and consistently. Not all birth control methods are equally effective. Female subjects of childbearing potential must use barrier contraception or hormonal contraception (such as oral contraceptives) to ensure that pregnancy does not occur.
12. The subjects are willing and able to comply with the schedule of visits, treatment plans, laboratory tests, and other requirements of the study.

Exclusion Criteria:

1. Suffering from other active malignant tumors within 3 years before randomization, except locally curable tumor types and those who have been cured, such as Squamous cell carcinoma of the skin, basal cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the breast.
2. Severe immunotherapy-related toxicity occurred during the previous anti-PD-1/PD-L1 monoclonal antibody treatment, including but not limited to: grade 3/4 pneumonia, proteinuria, uveitis or episcleritis, myasthenia gravis, Pancreatitis, hepatitis, bullous skin disease (including SJS, TEN); grade 2-4 encephalitis, myocarditis; any grade of Guillain-Barré syndrome, transverse myelitis; severe inflammation that significantly affects the quality of life of the patient sex joints.
3. Received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy, or other unmarketed clinical research drugs and other anti-tumor treatments within 4 weeks before the first use of the study drug.
4. Received nab-paclitaxel drug therapy within 6 months before the first use of the study drug. Known contraindications to nab-paclitaxel or hypersensitivity to any of its components.
5. Received drugs with immunomodulatory effects (such as thymosin, interferon, interleukin-2) within 2 weeks before randomization; received Chinese patent medicines with anti-tumor indications (such as Aidi injection, etc.) within 2 weeks before randomization.
6. Received major organ surgery (not including needle biopsy, etc.) or experienced significant trauma within 4 weeks before the first use of the study drug, or required elective surgery during the trial
7. There is central nervous system metastasis or cancerous meningitis.
8. Pleural effusion, pericardial effusion, or peritoneal effusion with uncontrollable need for repeated drainage (more than once a month) of subjects.
9. Suffering from active or recurrent autoimmune diseases; except the following: vitiligo, alopecia, psoriasis, or eczema that do not require systemic treatment; hypothyroidism caused by autoimmune thyroiditis that only requires stable doses of Hormone replacement therapy; type 1 diabetes requiring only a steady dose of insulin replacement therapy.
10. Subjects who need to use > 10 mg/day prednisone or equivalent dose of glucocorticoid or other immunosuppressive drugs for systemic treatment within 14 days before randomization; except the following

    1. Inhaled, ophthalmic or topical glucocorticoid therapy with a dose of ≤ 10 mg/day prednisone or equivalent dose is allowed.
    2. Physiological glucocorticoid replacement therapy, with a dose of ≤ 10 mg/day prednisone or an equivalent dose of glucocorticoid.
    3. Glucocorticoids as prophylaxis for hypersensitivity reactions (eg, before CT examination).
11. Live vaccines have been used within 4 weeks before randomization.
12. Known primary or secondary immunodeficiency, including human immunodeficiency virus (HIV) antibody test positive.
13. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
14. Known history of interstitial lung disease or non-infectious pneumonia.
15. Serious infection occurred within 4 weeks before randomization, including but not limited to complications requiring hospitalization, sepsis or severe pneumonia.
16. There are active infections that require systemic treatment (including active tuberculosis and active Treponema pallidum infection), and have used systemic antibacterial, antiviral or antifungal drugs within 2 weeks before randomization; Note: for type B Antiviral drugs used for viral hepatitis are excluded.
17. Active hepatitis B subjects, inactive or asymptomatic hepatitis B virus (HBV) carriers (hepatitis B surface antigen [HBsAg] positive) and HBV DNA> 1000 IU/mL), and subjects with active hepatitis C virus.
18. Suffering from active or documented inflammatory bowel disease (such as Crohn's disease, ulcerative colitis), active diverticulitis. There are clinical manifestations of gastrointestinal obstruction, or routine parenteral fluid rehydration, parenteral nutrition, or indwelling gastric tube are required.
19. Any of the following cardiovascular and cerebrovascular diseases:

    1. Myocardial infarction, unstable angina, pulmonary embolism, aortic dissection, deep venous thrombosis and any arterial thromboembolic events occurred within 6 months before randomization;
    2. Heart failure with New York Heart Association (NYHA) functional class ≥ II;
    3. There are severe arrhythmias that require long-term drug intervention; patients with atrial fibrillation who are asymptomatic and have stable ventricular rates are allowed;
    4. Cerebrovascular events (CVA) occurred within 6 months before randomization;
    5. Left ventricular ejection fraction (LVEF) < 50%;
    6. Previous history of myocarditis or cardiomyopathy.
    7. Hypertension (defined as systolic blood pressure > 150 mmHg, diastolic blood pressure > 100 mmHg) that remains uncontrolled after adequate antihypertensive drug treatment, or a history of hypertensive crisis or hypertensive encephalopathy.

       20) Known history of severe hypersensitivity to other monoclonal antibodies. 21) NCI CTCAE v5.0 ≥ grade 3 peripheral neuropathy exists. 22) The toxicity of previous anti-tumor therapy has not been relieved, defined as the toxicity has not recovered to NCI CTCAE v5.0 ≤ 2 grades, or the level specified in the inclusion/exclusion criteria (except hair loss) 23) The investigator believes that it may lead to risk of receiving the study drug treatment, or any condition that will interfere with the evaluation of the study drug or the safety of the subjects or the interpretation of the study results (such as suffering from other serious diseases or mental diseases, etc.).

       24) Enroll in another clinical study at the same time, unless it is an observational, non-interventional clinical study or follow-up period of an interventional study.

       25) Pregnant or lactating women. 26) Subjects considered by the investigator to be inappropriate to participate in the trial due to other reasons.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  To evaluate the clinical activity (as assessed by objective response rate [ORR]) of specific Cadonilimab and Nab-Paclitaxel combination.

SECONDARY OUTCOMES:
Duration of response | up to 2 years
  To evaluate the clinical activity (as assessed by duration of response (DoR)) of Cadonilimab and Nab-Paclitaxel combinations. DOR: length of time tumor continues to respond to the treatment.
Disease control rate (DCR) | up to 2 years
  Defined as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease.
Time to response (TTR) | up to 2 years
  Defined as the time from randomization to the date of the first confirmed documented response (CR or PR)
Progression Free survival | up to 2 years
  To evaluate the clinical activity (as assessed by progression-free survival [PFS]) of Cadonilimab and Nab-Paclitaxel combinations. PFS: Time from treatment initiation to the first documented disease progression per response evaluation criteria in solid tumors (RECIST) 1.1 as assessed by local site or death, whichever occurs first.
Overall survival | Cycle 1 Day 1, Day 1 of each cycle (each cycle is 21 days), every 12 weeks after end of treatment
  To evaluate the clinical activity (as assessed by overall survival [OS]) of Cadonilimab and Nab-Paclitaxel combinations. OS: Time from treatment initiation to death due to any cause.
Incidence of adverse events | Day 1 of each cycle (each cycle is 21 days), up to 2 years
  To evaluate the safety and tolerability of Cadonilimab and Nab-Paclitaxel combination:
  Number of Participants Experiencing Adverse Events (AEs) according to NCI CTCAE Version 5.0.
Health-Related Quality of Life (HRQoL) Assessed by European Organisation for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 (QLQC30) Score | At baseline (prior to first dose of study drug), on Day 1 of each subsequent cycle (cycle length of 21 days), and at the post-treatment visit (up to 2 years)
  EORTC QLQ-C30 was a questionnaire which included 30 questions that rates the overall quality of life in cancer participants. The first 28 questions use a 4-point scale (1=not at all to 4=very much) for evaluating function (physical, role, social, cognitive, emotional), symptoms (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea/vomiting, constipation, and pain) and financial difficulties. The last 2 questions use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Scores are transformed to a range of 0 to 100 using a standard EORTC algorithm. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/quality of life (QoL) represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problem.

OTHER OUTCOMES:
Exploratory endpoints | Within 7 days before treatment, 6 weeks ± 7 days after treatment, 12 weeks ± 7 days after treatment
  Evaluate the correlation between therapeutic effect and immune cells (T cells, B cells, myeloid and other subgroups), TCR, HPV, cytokines in tumor tissue and peripheral blood, and analyze the immune-resistant microenvironment characteristics, Dynamic changes of immune microenvironment before and after treatment with cadonilimab combined with nab-paclitaxel. Genomic profile predicts efficacy of cadonilimab combined with Nab-Paclitaxel.

CONTACTS AND LOCATIONS:
Overall Officials: hui Wang, PHD, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University; bairong xia, PHD, Principal Investigator — Anhui Provincial Cancer Hospital; Ge Lou, PHD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University